CLINICAL TRIAL: NCT01909986
Title: An Open Label, Single-dose Study to Evaluate the Pharmacokinetics, Metabolism and Excretion Balance of [14C]-ONO-4053 in Healthy Adult Male Subjects
Brief Title: A Human Mass Balance Study to Determine the Total Recovery of Radioactivity in Urine and Faeces Following a Single Oral Dose of 14C Radiolabelled ONO-4053
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ONO-4053POE004
Record Dates: First submitted 2013-07-08; First posted 2013-07-29 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Adult Male Subjects
Keywords: ONO-4053; Healthy adult male subjects; pharmacokinetics; metabolism; excretion; mass balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E1 (Experimental): [14C]-ONO-4053
  Interventions: Drug: [14C]ONO-4053

INTERVENTIONS:
Drug: [14C]ONO-4053 — Single dose [14C]ONO-4053

SUMMARY:
This is a single dose mass balance study in healthy adult male volunteers to investigate the metabolism and excretion of [14C]-ONO-4053.

DETAILED DESCRIPTION:
This is a single centre, open-label, non-randomised study in healthy adult male subjects. Six subjects will receive a single dose of 14C ONO-4053 administered orally as a suspension. Safety measurements (ECG, vital signs, biochemistry and haematology) and adverse events will be monitored throughout the study. After administration of 14C ONO-4053 subjects will remain in the clinical facility for collection of blood, urine and faecessamples. Samples will be analysed for recovery of radioactivity and characterisation of metabolites of ONO-4053.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent
2. Healthy male subjects aged 35 to 65 years inclusive
3. Subject is not trying to father a child and is willing to use one of the contraception methods listed in the protocol 4 The subject has a body mass index of 19.0 to 30.0 kg/m2 inclusive. 5 The subject is healthy as determined by the Investigator 6 Regular daily bowel movements

Exclusion Criteria:

1. The Investigator deems the subject unsuitable for the study
2. The subject has, or has a history of, any significant disease or disorder (including any clinically significant laboratory findings) that would increase the risk for the subject if they were enrolled in the study
3. The subject has a history of acute gastrointestinal illness
4. The subject has used prescription medicine, non-prescription medicine, vitamins, herbal treatments or dietary supplements within 14 days of dosing.
5. Current smokers and those who have smoked within the last 12 months
6. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
[14C]ONO-4053 recovery | 11 Days
  Total recovery of radioactivity in urine and faeces expressed as a percentage of the total radioactive dose administered

SECONDARY OUTCOMES:
[14C]-ONO-4053 metabolites | 11 Days
  Characterisation and identification of [14C]-ONO-4053 metabolites in plasma, urine and faeces.
Total drug-related material | 11 Days
  PK parameters of total drug-related material (radioactivity) in blood and plasma
ONO-4053 in plasma | 11 Days
  PK parameters of ONO-4053 in plasma
Blood:plasma ratio of [14C]ONO-4053 | 11 Days
  Blood:plasma ratio of total drug-related material (radioactivity)
Radioactivity in urine | 11 Days
  PK parameter of total radioactivity in urine
Safety and tolerability parameters | 14 - 16 days
  Safety and tolerability parameters including collection of adverse events, physical examinations, vital signs, 12-Lead ECG and laboratory evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Nottingham Clinical site, Nottingham, United Kingdom